CLINICAL TRIAL: NCT03357250
Title: Validation of Biomarkers of Adverse Neurologic Outcome in Newborns Who Required Resuscitation or Are Suspected to be at Risk for Perinatal Brain Injury and Long-term Adverse Neurological Outcome A Prospective Multicenter Observational Study for Development of a Diagnostic Test
Brief Title: Biomarkers And Neurological Outcome in Neonates (BANON)
Status: Completed | Type: Observational
Sponsor: Life Science Inkubator (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: BANON I
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-11

CONDITIONS: Asphyxia Neonatorum
Keywords: biomarkers
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples Without DNA — blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Validation of biomarkers in a human population for their ability to diagnose the severity of neonatal asphyxia. These biomarkers linked to asphyxia have been identified in animal studies and a preliminary human study.

DETAILED DESCRIPTION:
The aim of the study is to validate the application of combinations of several laboratory parameters in early postnatal blood samples, for identification of infants, who will suffer from early abnormal neonatal neurological outcome, in a population at risk.

The population at risk is defined as term and late preterm (>36 weeks of gestation) human infants following perinatal hypoxia-ischemia with or without postnatal resuscitation, and where the combination of laboratory parameters is derived from a preliminary study performed in Turkey (AAMBI) using a metabolomics approach.

ELIGIBILITY:
Inclusion Criteria:

* Need for resuscitation after birth: For >1 min. after birth, positive pressure respiratory support with face mask or endotracheal tube (but not only CPAP), or cardiac compressions
* 5 min APGAR-score ≤ 5.
* Perinatal hypoxia-ischemia defined as a perinatal acidosis indicated by a pH≤7.1 in arterial umbilical cord blood or early postnatal blood collected at <30min of age
* Perinatal hypoxia-ischemia indicated by a base deficit ≥ 12mmol/l in umbilical cord blood or early postnatal blood collected at <30min of age.

Exclusion Criteria:

* Age >1.5h
* gestational age < 36 weeks
* birth weight <2000g
* congenital malformation
* missing valid written informed parental consent
* unsuccessful resuscitation
* infant considered not-viable
* decision for palliative care only

Ages: 0 Minutes to 90 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants at risk for perinatal hypoxic-ischemic brain injury
Sampling Method: Probability Sample
Enrollment: 553 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Validation of diagnostic algorithm | 10 days
  The best combinations of biomarkers from the preliminary study will be used and sensitivity and specificity as well as positive and negative likelihood ratios and their 95%-confidence limits will be calculated.

CONTACTS AND LOCATIONS:
Locations (11):
- Germany (11):
  - Abt. Neonatologie und Päd. Intensivmedizin Klinikum, Aschaffenburg
  - Neonatologie Universitätsklinikum, Dresden
  - Universitätsklinikum Essen Klinik für Kinderheilkunde I Neonatologie, Essen
  - Marienkrankenhaus im Wilhelmstift, Hamburg
  - Universitätsklinikum Heidelberg Neonatologie, Heidelberg
  - Klinik für Kinder- und Jugendmedizin, Karlsruhe
  - Klinik für Kinder- und Jugendmedizin, Klinikum Dritter Orden, München
  - Haunersches Kinderspital am Perinatalzentrum Grosshadern, München
  - Kinderklinik Dritter Orden, Passau
  - Klinik St. Hedwig Neonatologie, Regensburg
  - Klinik für Kinder und Jugendmedizin, Tübingen

IPD SHARING:
Plan to Share IPD: No